CLINICAL TRIAL: NCT01832402
Title: A Preliminary Study of Prophylactic Fentanyl Pectin Nasal Spray (FPNS) for Exercise-Induced Breakthrough Dyspnea
Brief Title: Fentanyl Pectin Nasal Spray (FNPS) for Exercise-Induced Breakthrough Dyspnea
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: Depomed (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: 2012-1169; NCI-2013-00961 (Registry Identifier: NCI CTRP)
Record Dates: First submitted 2013-04-10; First posted 2013-04-16 (Estimated); Results first posted 2020-09-04 (Actual); Last update posted 2023-06-08 (Actual); Status verified 2023-06

CONDITIONS: Advanced Cancers
Keywords: Advanced Cancers; Exercise-Induced Breakthrough Dyspnea; Shortness of breath; Fentanyl pectin nasal spray; Placebo nasal spray; Walk test; Questionnaires; Surveys; Mental ability tests
MeSH Terms: conditions — Dyspnea | interventions — Surveys and Questionnaires

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Fentanyl Pectin Nasal Spray (Experimental): Fentanyl pectin nasal (FPNS) dose equivalent to 15-25% of the morphine equivalent daily dose (MEDD). FPNS administered intranasally 20 minutes before the second 6-minute walk test. Same dose repeated at least 30 minutes after the first dose and 20 minutes prior to the third and final 6 minute walk test. Walk test administered before first dose of FPNS. Participant will rest for 30 minutes after walk test. FPNS administered, then participant will wait 20 minutes before repeating second 6 minute walk test. After second walk test, participant will rest for 30 minutes. FPNS administered for second time, then participant will wait for 20 minutes. Walk test administered again for 6 minutes. Questionnaires completed at baseline, before each walk test, and at end of final walk test. Four mental ability tests administered after each walk test to include finger tapping, simple mathematics questions, recall of numbers, and recall of objects.
  Interventions: Drug: Fentanyl Pectin Nasal Spray; Other: Walk Test; Behavioral: Questionnaires; Behavioral: Mental Ability Tests
- Placebo Nasal Spray (Placebo Comparator): Placebo nasal spray administered intranasally 20 minutes before the second 6-minute walk test. Same dose repeated at least 30 minutes after the first dose and 20 minutes prior to the third and final 6 minute walk test. Walk test administered before first dose of placebo nasal spray. Participant will rest for 30 minutes after walk test. Placebo nasal spray administered, then participant will wait 20 minutes before repeating second 6 minute walk test. After second walk test, participant will rest for 30 minutes. Placebo nasal spray administered for second time, then participant will wait for 20 minutes. Walk test administered again for 6 minutes. Questionnaires completed at baseline, before each walk test, and at end of final walk test. Four mental ability tests administered after each walk test to include finger tapping, simple mathematics questions, recall of numbers, and recall of objects.
  Interventions: Drug: Placebo Nasal Spray; Other: Walk Test; Behavioral: Questionnaires; Behavioral: Mental Ability Tests

INTERVENTIONS:
Drug: Fentanyl Pectin Nasal Spray — Fentanyl pectin nasal (FPNS) dose equivalent to 15-25% of the morphine equivalent daily dose (MEDD) administered intranasally 20 minutes before the second 6-minute walk test. Same dose repeated at least 30 minutes after the first dose and 20 minutes prior to the third and final 6 minute walk test.
  Arms: Fentanyl Pectin Nasal Spray
Drug: Placebo Nasal Spray — Placebo nasal spray administered intranasally 20 minutes before the second 6-minute walk test. Same dose repeated at least 30 minutes after the first dose and 20 minutes prior to the third and final 6 minute walk test.
  Arms: Placebo Nasal Spray
Other: Walk Test — Walk test administered before first dose of drug/placebo nasal spray. Participant will rest for 30 minutes after walk test. Drug/placebo nasal spray administered, then participant will wait 20 minutes before repeating second 6 minute walk test. After second walk test, participant will rest for 30 minutes. Drug/placebo nasal spray administered for second time, then participant will wait for 20 minutes. Walk test administered again for 6 minutes.
Behavioral: Questionnaires — Questionnaires completed at baseline, before each walk test, and at end of final walk test.
  Other Names: Surveys
Behavioral: Mental Ability Tests — Four mental ability tests administered after each walk test to include finger tapping, simple mathematics questions, recall of numbers, and recall of objects.

SUMMARY:
The goal of this clinical research study is to learn if fentanyl nasal spray can help to control shortness of breath in patients who have been treated or are being treated for cancer.

Fentanyl is commonly used for treatment of cancer pain. It may help patients with their shortness of breath as well.

In this study, fentanyl will be compared to a placebo. A placebo is not a drug. It looks like the study drug but is not designed to treat any disease or illness. It is designed to be compared with a study drug to learn if the study drug has any real effect.

DETAILED DESCRIPTION:
Study Groups:

If you are found to be eligible to take part in this study, you will be randomly assigned (as in the flip of a coin) to receive either fentanyl or placebo. You will have an equal chance of being assigned to either group. Neither you nor the study staff will know to which group you have been assigned. However, if needed for your safety, the study staff will be able to find out what you are receiving.

Study Drug/Placebo Administration:

Before you receive the study drug/placebo, you will walk back and forth in an indoor hallway for up to 6 minutes. You may feel out of breath or become exhausted. You may slow down, stop, and rest at any time you need to.

After that, you will sit down and rest (for about 30 minutes).

You will then be given the study drug/placebo by a nasal spray. You will then wait for another 20 minutes and repeat the walking test.

After that, you will sit down and rest (for about 30 minutes).

You will then be given the study drug/placebo again by a nasal spray. You will then wait for another 20 minutes and repeat the walking test for a third time.

Study Visit:

During your study visit, the study staff will collect information from your medical record about your age, sex, race, disease type, your performance status, any drugs you are taking, and possible causes of shortness of breath.

Before each walk test, you will complete the questionnaires about your symptoms.

Before and after each walk test, the study staff will record your heart rate, breathing rate, and the level of oxygen in your blood using a measuring device that will be clipped onto your finger. The study staff will also ask you 3 questions about how hard it is to catch your breath and your level of tiredness.

During each walk test, you will be asked 6 times how hard it is to catch your breath. The distance you walked and how often and for how long you stopped will be recorded.

Before and after the second and third walk tests, the study staff will ask you about any side effects from the study drug/placebo that you may be having.

During the rest period between the walk tests, you may be asked several times how hard it is to catch your breath.

After each walk test, you will also be asked to complete 4 tests of your mental abilities, including finger tapping, simple mathematics questions (addition, subtraction, multiplication, division), recall of numbers, and recall of objects. It should take 15 minutes to complete these tests.

At the end of the study visit, you will complete 1 questionnaire that asks if you think the study drug/placebo is helping you, and how satisfied you are with the study. It should take about 5 minutes to complete the questionnaire.

Length of Study:

You will be on this study for up to 3 hours. You will be taken off study if intolerable side effects occur during the study.

This is an investigational study. Fentanyl is FDA approved and commercially available for the treatment of pain. Its use to help with shortness of breath is investigational.

Up to 25 patients will be enrolled in this study. All will be enrolled at MD Anderson.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosis of cancer
2. Breakthrough dyspnea, defined in this study as dyspnea on exertion with an average intensity level >=3/10 on the numeric rating scale
3. Outpatient at MD Anderson Cancer Center seen by the Supportive Care Service or Thoracic Medical Oncology
4. Ambulatory and able to walk with or without walking aid
5. On strong opioids with morphine equivalent daily dose of 80-500 mg, with stable (i.e. +/- 30%) regular dose over the last 24 hours
6. Karnofsky performance status >=50%
7. Age 18 or older
8. Able to complete study assessments

Exclusion Criteria:

1. Dyspnea at rest >=7/10 at the time of enrollment
2. Supplemental oxygen requirement >6 L per minute
3. Delirium (i.e. Memorial delirium rating scale >13)
4. History of unstable angina or myocardial infarction 1 month prior to study enrollment
5. Resting heart rate >120 at the time of study enrollment
6. Systolic pressure >180 mmHg or diastolic pressure >100 mmHg at the time of study enrollment
7. History of active opioid abuse within the past 12 months
8. History of allergy to fentanyl
9. Unwilling to provide informed consent
10. Patients who currently have no evidence of disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Actual)
Dates: Start 2013-06-11 (Actual); Primary Completion 2019-11-25 (Actual); Study Completion 2019-11-25 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David Hui, MD, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- University of Texas MD Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- [Derived] Hui D, Kilgore K, Park M, Williams J, Liu D, Bruera E. Impact of Prophylactic Fentanyl Pectin Nasal Spray on Exercise-Induced Episodic Dyspnea in Cancer Patients: A Double-Blind, Randomized Controlled Trial. J Pain Symptom Manage. 2016 Oct;52(4):459-468.e1. doi: 10.1016/j.jpainsymman.2016.05.013. Epub 2016 Jul 9. PMID 27401508
- See also: University of Texas MD Anderson Cancer Center Website — http://www.mdanderson.org

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Adult participants (age>18) with an active diagnosis of cancer were recruited between 6/2013 and 3/2015 from the Supportive Care Center outpatient clinic of MD Anderson Cancer Center who satisfied the inclusion and exclusion criteria.
Groups:
- Intervention Group (Fentanyl Pectin Nasal Spray): Received Fentanyl Pectin Nasal Spray 20 minutes before 2nd and 3rd 6 minute walk tests, dose equivalent to 15-25% of total daily opioid dose each time.
- Controlled Group (Placebo): Received similar number of Placebo Spray 20 minutes before 2nd and 3rd 6 minute walk tests.
Period: Overall Study
Arm/Group | Intervention Group (Fentanyl Pectin Nasal Spray) | Controlled Group (Placebo)
Started | 19 | 16
Received Allocated Medication | 12 | 12
Completed Study With Correct Dose | 10 | 9
Completed Study With Incorrect Dose | 2 | 3
Completed | 12 | 12
Not Completed | 7 | 4
Not completed — Lost to Follow-up | 2 | 0
Not completed — Withdrawal by Subject | 3 | 3
Not completed — Declining Performance status | 2 | 1

BASELINE CHARACTERISTICS:
Population: Intention to treat analysis participants data
Groups:
- Total: Total of all reporting groups
Arm/Group | Intervention Group (Fentanyl Pectin Nasal Spray) | Controlled Group (Placebo) | Total
Number analyzed (Participants) | 12 | 12 | 24
Age, Continuous [Mean (Inter-Quartile Range); unit: Years] | 51.5 [44.7 to 58.3] | 53.3 [45.0 to 61.6] | 52.4 [47.5 to 57.4]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9 | 4 | 13
  Male | 3 | 8 | 11
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 2 | 3
  Not Hispanic or Latino | 11 | 10 | 21
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 3 | 2 | 5
  White | 9 | 10 | 19
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 12 | 12 | 24
Education [Count of Participants; unit: Participants]
  High School or less | 4 | 2 | 6
  College | 8 | 7 | 15
  Advanced Degree | 0 | 3 | 3
Cancer Type [Count of Participants; unit: Participants]
  GastroIntestinal Cancer | 2 | 4 | 6
  Breast Cancer | 3 | 2 | 5
  Lung Cancer | 1 | 2 | 3
  Genitourinary Cancer | 2 | 0 | 2
  Gynecologic Cancer | 2 | 0 | 2
  Hematologic | 0 | 2 | 2
  Others | 2 | 2 | 4
Cancer Stage [Count of Participants; unit: Participants]
  Metastatic Stage | 8 | 10 | 18
  Localized/Locally advanced | 4 | 2 | 6
Comorbidity [Count of Participants; unit: Participants]
  Asthma | 5 | 0 | 5
  COPD | 2 | 2 | 4
  Heart Failure | 1 | 0 | 1

OUTCOME MEASURES:

1. Primary Outcome: Dyspnea Numeric Rating Scale
Description: Our primary outcome was dyspnea intensity "now" using a dyspnea numeric rating scale that ranges from 0 ("no shortness of breath") to 10 ("worst possible shortness of breath"). Measured the mean difference of dyspnea numeric rating scale between the first and second 6 Minute Walk Tests and between the first and third 6 Minute Walk Tests. 6 minute walk tests were carried out following guidelines from the American Thoracic Society.
Time Frame: 1.5 to 2 hours on a Single visit
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Intervention Group (Fentanyl Pectin Nasal Spray) | Controlled Group (Placebo)
Number analyzed (Participants) | 12 | 12
score on a scale
  Mean difference between 1st and 2nd walk tests | -2.0 [-3.5 to -0.6] | -1.7 [-3.3 to -0.1]
  Mean difference between 1st and 3rd walk tests | -2.3 [-4.0 to -0.7] | -2.5 [-4.2 to -0.9]

2. Secondary Outcome: Dyspnea Borg Scale
Description: Assessed dyspnea using the modified Dyspnea Borg Scale that ranges from 0 ("no shortness of breath") to 10 ("worst possible shortness of breath"). Measured the mean difference of modified Dyspnea Borg scale between the first and second 6 Minute Walk Tests and between the first and third 6 Minute Walk Tests.
Time Frame: 1.5 to 2 hours on a Single visit
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Intervention Group (Fentanyl Pectin Nasal Spray) | Controlled Group (Placebo)
Number analyzed (Participants) | 12 | 12
score on a scale
  Mean difference between 1st and 2nd walk tests | -1.8 [-3.1 to -0.4] | -1.7 [-3.3 to -0.1]
  Mean difference between 1st and 3rd walk tests | -1.7 [-3.5 to 0] | -2.4 [-4.2 to -0.6]

3. Secondary Outcome: Walk Distance at 6 Minutes
Description: Compared the mean difference of distance between the first and second 6 Minute Walk Tests and between the first and third 6 Minute Walk Tests.
Time Frame: 1.5 to 2 hours on a Single visit
Measure: Mean (95% Confidence Interval); unit: meters
Groups:
- Interventional Group (Fentanyl Pectin Nasal Spray): Received Fentanyl Pectin Nasal Spray 20 minutes before 2nd and 3rd 6 minute walk tests, dose equivalent to 15-25% of total daily opioid dose each time.
- Control Group (Placebo): Received similar number of Placebo Spray 20 minutes before 2nd and 3rd 6 minute walk tests.
Arm/Group | Interventional Group (Fentanyl Pectin Nasal Spray) | Control Group (Placebo)
Number analyzed (Participants) | 12 | 12
meters
  Mean difference between 1st and 2nd walk tests | 23.8 [1.3 to 46.2] | 16.3 [-8.6 to 41.3]
  Mean difference between 1st and 3rd walk tests | 23.3 [-1.7 to 48.2] | 14.6 [-11.0 to 40.3]

ADVERSE EVENTS:
Time Frame: Baseline, up to 2 hours in one single visit
Description: Each adverse effect was measured using an 11-point numeric rating scale (0=none, 10=worst) before drug administration and immediately after the 2nd 6 minute walk test (approximately 30 minutes later) and immediately again after the 3rd 6 minute walk test (again measured approximately 30 minutes later).
Groups:
- Interventional (Fentanyl Pectin Nasal Spray) Second Walk Test: Received Fentanyl Pectin Nasal Spray 20 minutes before 2nd 6 minute walk tests, dose equivalent to 15-25% of total daily opioid dose each time.
- Control (Placebo), Second Walk Test: Received similar number of Placebo Spray 20 minutes before 2nd 6 minute walk tests.
- Interventional (Fentanyl Pectin Nasal Spray),Third Walk Test: Received Fentanyl Pectin Nasal Spray 20 minutes before 3rd 6 minute walk tests, dose equivalent to 15-25% of total daily opioid dose each time.
- Control (Placebo), Third Walk Test: Received similar Placebo Spray 20 minutes before 3rd 6 minute walk tests.
Arm/Group | Interventional (Fentanyl Pectin Nasal Spray) Second Walk Test | Control (Placebo), Second Walk Test | Interventional (Fentanyl Pectin Nasal Spray),Third Walk Test | Control (Placebo), Third Walk Test
All-Cause Mortality (participants affected / at risk) | 0/12 | 0/12 | 0/12 | 0/12
Serious Adverse Events (participants affected / at risk) | 0/12 | 0/12 | 0/12 | 0/12
Other Adverse Events (participants affected / at risk) | 2/12 | 2/12 | 5/12 | 5/12
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Interventional (Fentanyl Pectin Nasal Spray) Second Walk Test (N=12) | Control (Placebo), Second Walk Test (N=12) | Interventional (Fentanyl Pectin Nasal Spray),Third Walk Test (N=12) | Control (Placebo), Third Walk Test (N=12)
Nausea (Gastrointestinal disorders) | 0 | 0 | 2 | 0
Dizziness (Nervous system disorders) | 2 | 2 | 5 | 1
Drowsiness (Nervous system disorders) | 1 | 2 | 1 | 5
Stuffy Nose (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 0 | 0
Nose Dryness (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 0 | 2
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 1
Sore throat (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2013-11-05): https://cdn.clinicaltrials.gov/large-docs/02/NCT01832402/Prot_SAP_000.pdf